CLINICAL TRIAL: NCT06407453
Title: Effectiveness of Exercise Given With Ergonomics Training in Tea Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar6
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain; Back Pain; Work-related Illness
MeSH Terms: conditions — Neck Pain; Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): No intervention will be made
  Interventions: Other: control
- exercise (Experimental): exercise program will be applied
  Interventions: Other: exercise

INTERVENTIONS:
Other: control — There will be no interference ergonomics training
  Arms: control
Other: exercise — upper extremity strengthening exercises upper extremity stretching exercises ergonomics training posture training relaxation exercises
  Arms: exercise

SUMMARY:
The aim of our study is to investigate the effectiveness of exercise against work-related musculoskeletal disorders in tea workers.

DETAILED DESCRIPTION:
Individuals who volunteer to participate in the study will be evaluated considering the inclusion and exclusion criteria, and participants will participate in the study after reading and signing the Informed Consent Form. Tea workers who collect tea will be divided into 2 groups. .Demographic Information Form, Visual Analogue Scale (VAS), Upper Extremity Discomfort Analysis, Rapid Upper Extremity Assessment (RULA), Sleep Quality, Scandinavian Musculoskeletal System Questionnaire will be given to the participants of both groups. The surveys will be carried out face to face. After the application of the surveys, statistical data will be obtained. analyzes will be made. One group will be given exercise, the other group will not be given exercise. Post-exercise surveys will be conducted again to check the effectiveness of the exercise.

ELIGIBILITY:
INCLUSION CRITERIA

* Being between the ages of 25-45.
* Having been a tea craftsman for at least 10 years.
* Having the ability to read and write Turkish.
* Agreeing to participate in the study voluntarily.

EXCLUSION CRITERIA

* Being diagnosed with a serious psychological illness.
* Malignancy
* Advanced osteoporosis
* Being under 25 years of age.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Arm Shoulder and Hand Problems Questionnaire | 14 weeks
  It is a questionnaire developed by the American Academy of Orthopedic Surgeons (AAOS) based on the World Health Organization (WHO) model and used to evaluate upper extremity function status. The survey consists of three parts, and for all questions in the scale, the person marks the answer that suits him or her on a 5-point Likert system (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: not able to do it at all). According to the results of the Arm Shoulder and Hand Problems Questionnaire survey; A result between 0-100 is obtained from each section (0: no problem, 100: maximum problem).
Nordic Musculoskeletal Survey | 14 weeks
  It consists of 11 questions asked as a reference from 9 body regions shown on a visual body diagram of neck, shoulder, back, elbow, hand, wrist, waist, hip, thigh, knee, foot, ankle, and corresponds to 99 data items. The questionnaire primarily questions the presence of pain in 9 body regions. If the person's answer is yes, he moves on to the relevant sub-questions.It is a selection scale rather than a rating.
Pittsburgh Sleep Quality Index | 14 weeks
  The scale is a 19-item self-report scale that evaluates sleep quality and disturbance over the past month. It consists of 24 questions, 19 questions are self-report questions, 5 questions are questions to be answered by the spouse or roommate. The 18 scored questions of the scale consist of 7 components. Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disturbance, Sleeping Medication Use, and Daytime Dysfunction. Each component is evaluated on a scale of 0-3 points. The total score of the 7 components gives the scale total score. Total score varies between 0-21. A total score greater than 5 indicates "poor sleep quality".

CONTACTS AND LOCATIONS:
Overall Officials: İlayda GÜR, Study Chair — Uskudar University
Locations (1):
- Uskudar Üniversity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhattacharyya N, Chakrabarti D. Ergonomic basket design to reduce cumulative trauma disorders in tea leaf plucking operation. Work. 2012;41 Suppl 1:1234-8. doi: 10.3233/WOR-2012-0308-1234. PMID 22316888
- [Background] Mirbod SM, Fujita S, Miyashita K, Inaba R, Iwata H. Some aspects of occupational safety and health in green tea workers. Ind Health. 1995;33(3):101-17. doi: 10.2486/indhealth.33.101. PMID 8543474
- [Background] Lallukka T, Hiilamo A, Oakman J, Manty M, Pietilainen O, Rahkonen O, Kouvonen A, Halonen JI. Recurrent pain and work disability: a record linkage study. Int Arch Occup Environ Health. 2020 May;93(4):421-432. doi: 10.1007/s00420-019-01494-5. Epub 2019 Nov 28. PMID 31781902
- [Background] Marak TR, Bhagat D, Borah S. Musculoskeletal Disorders of Garo Women Workers Engaged in Tea-Plucking Activity: An Ergonomic Analysis. Indian J Occup Environ Med. 2020 May-Aug;24(2):60-65. doi: 10.4103/ijoem.IJOEM_185_19. Epub 2020 Aug 19. PMID 33281373
- [Background] Kairi TK, Dey S. Prevalence of work-related musculoskeletal symptoms among tea garden workers in Bangladesh: a cross-sectional study. BMJ Open. 2022 May 9;12(5):e061305. doi: 10.1136/bmjopen-2022-061305. PMID 35534079
- [Derived] Gur I, Sevgin O, Dikmen Hosbas B. Effectiveness of ergonomics training and exercise in tea workers: a randomized controlled trial. Int Arch Occup Environ Health. 2025 Dec;98(9-10):945-955. doi: 10.1007/s00420-025-02185-0. Epub 2025 Nov 18. PMID 41251731